CLINICAL TRIAL: NCT00300573
Title: A Randomized, Double-Blind, Phase II Study Comparing the Anti-Retroviral Safety and Efficacy of Dexelvucitabine (DFC) 200 mg Once Daily to Lamivudine (3TC) 300 mg Once Daily in Addition to Optimized Background Therapy in HIV-1 Infected Subjects Who Have Failed and/or Harbor HIV With Resistance Mutations to NRTIs, PIs, and NNRTIs
Brief Title: Randomized, Double-Blind Study Comparing Dexelvucitabine (DFC) to Lamivudine (3TC) in Subjects With Resistance to NRTIs, PIs, and NNRTIs
Acronym: DECLARE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development program ended due to inability to pair with other cytidine analogs and higher risk of hyperlipasemia when not used with 3TC/FTC.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 08721-204; EudraCT #:2006-000096-16
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections; Human Immunodeficiency Virus
Keywords: dexelvucitabine; DFC; Treatment Experienced; HIV-1
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — dexelvucitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexelvucitabine (DFC) (Experimental): 200 mg once daily
  Interventions: Drug: Dexelvucitabine
- lamivudine (3TC) (Active Comparator): 300 mg once daily
  Interventions: Drug: Dexelvucitabine

INTERVENTIONS:
Drug: Dexelvucitabine — nucleoside inhibitor of HIV Reverse Transcriptase

SUMMARY:
The study will compare the safety and efficacy of an investigation nucleoside analog reverse transcriptase inhibitor (NRTI), dexelvucitabine (DFC), to an approved NRTI, lamivudine (3TC) in HIV treatment-experienced patients who are resistant to 3 classes of antiretroviral therapies (NRTIs, PIs and NNRTIs). Patients meeting eligibility requirements will have a new 'optimized' background regimen (OBR) selected for them by their investigator based on prior ARV treatment history and the results of HIV genotype and phenotype tests performed during the screening period. In addition to treatment with the new OBR, patients will be randomized to receive treatment with either DFC or 3TC in a blinded fashion. There is a 50 percent chance a patient will receive DFC or 3TC. Treatment in the study may continue for up to 96 weeks. Patients with an inadequate response to therapy after 16 weeks will have the option to change their OBR and the option to switch to receive the other study medication (i.e., DFC to 3TC or 3TC to DFC).

DETAILED DESCRIPTION:
The study will compare the safety and efficacy of an investigational nucleoside analog reverse transcriptase inhibitor (NRTI), dexelvucitabine (DFC) 200 mg once daily, to an approved NRTI, lamivudine (3TC) 300 mg once daily in treatment experienced patients with HIV that is resistant to 3 classes of antiretroviral therapies (NRTIs, PIs and NNRTIs). Patients meeting eligibility requirements will have a new 'optimized' background regimen (OBR) selected for them based on prior treatment history, and results of HIV genotype and phenotype performed during screening. In addition to the OBR patients will be randomized to receive at at one to one ratio DFC or 3TC in a blinded fashion. The OBR may include any approved HIV treatments except 3TC, FTC, ddI, d4T and ddC. Medications available through expanded access may also be available to selected patients. Treatment in the study will continue for up to 96 weeks with primary endpoints at 24 and 48 weeks of therapy. Patients with an inadequate response to therapy after 16 weeks will have the option to change their OBR and the option to switch study medication (DFC to 3TC or 3TC to DFC). A total of 250 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* a) Male (at birth) subjects, between 16 years (or the legal age of consent, whichever is older) and 75 years of age, utilizing adequate contraceptive methods.
* b) Female (at birth) subjects between 16 years (or the legal age of consent, whichever is older) and 75 years of age.
* Women of childbearing potential may be enrolled following a negative serum pregnancy test. If participating in activity that could lead to pregnancy, women shall agree to use TWO forms of contraception as listed in # 1-4 below (at least one must be a barrier method) while receiving protocol-specified medication and for 2 months after stopping the medication.

  1. Condom (male or female) with or without a spermicidal agent
  2. Diaphragm or cervical cap with spermicide
  3. IUD
  4. Hormonal-based contraception
* Women who are not of reproductive potential (documented to be surgically sterile or postmenopausal [defined as amenorrhea >1 year and follicle stimulating hormone {FSH} >30 mU/mL]) are eligible to be enrolled without a serum pregnancy test and will not be required to use contraception.
* Subjects treated with a HAART regimen(s), including a minimum of 3 drugs, for at least 3 months and who have been on a stable HAART regimen for a minimum of 8 weeks prior to the Screening visit. The HAART regimen must also remain stable from the Screening visit until randomization on Day 0 in order for the subject to qualify for enrollment.
* Demonstrate evidence of failure of at least 3 drug classes, defined as #s 1-3 below:

  1. Prior NRTI use and presence of one or more NRTI-resistance-conferring mutations, including mutations at RT amino acids 41L, 65R, 67N, 70R, 74V or 74I, 184V or 184I, 210W, 215Y or 215F, and/or 219Q or 219E.
  2. Presence of one or more NNRTI-resistance conferring mutations, including mutations at RT amino acids 100I, 101E or 101P, 103N, 106A or 106M, 188L, and/or 190A or 190S or 190E at Screening or documented to be present on a prior genotype OR documented evidence of prior NNRTI use of at least 2 months duration with viral load ≥1000 copies/mL after at least 2 months of treatment.
  3. Prior ritonavir-boosted PI use AND presence of one or more PI-resistance-conferring mutations, including mutations at protease amino acids 33F, 46I or 46L, 50V, 82A or 82F or 82T or 82S, 84V, and/or 90M.
* Demonstrate a Screening plasma HIV RNA concentration of ³1000 copies/mL (Roche Amplicor HIV-1 Monitor® Test, v1.5 - Quantitative assay) and, in the expert judgment of the investigator, be failing the current regimen.
* Be able and willing to provide written informed consent.
* Be able and willing to comply, in the opinion of the investigator, with the requirements of this study.

Exclusion Criteria:

* Current or recent (<30 days) opportunistic infection (Category C according to the Centers for Disease Control (CDC) Classification System for HIV-1 Infection, 1993 Revised Version) that is not being controlled by medication in the judgment of the investigator.
* Subjects who are, in the opinion of the investigator, unable to comply with the dosing schedule and protocol evaluations.
* Pregnant women or women who are breastfeeding
* Current alcohol or drug use, which in the expert judgment of the investigator, will interfere with the subject's ability to comply with the protocol requirements.
* Subjects treated with dexelvucitabine (formerly known as Reverset) in a prior investigational drug protocol.
* Subjects with a history of acute or chronic pancreatitis.
* Subjects with acute hepatitis B and/or C infection.
* Subjects with unstable chronic hepatitis.
* Subjects with chronic renal failure requiring dialysis.
* Subjects currently receiving 3TC or FTC as part of a regimen for treatment of stable, chronic HBV infection. Subjects with stable chronic HBV infection who are being treated with entecavir, adefovir, or tenofovir are eligible to enroll.
* Subjects with the following laboratory parameters within 35 days prior to first dose of study medication:

  * Hemoglobin <9.0 g/dL (males) or <8.0 g/dL (females)
  * Absolute neutrophil count (ANC) <750/mm3
  * Platelet count <75 000/mm3
  * Aspartate aminotransaminase (AST [SGOT]) or alanine aminotransaminase (ALT [SGPT]) >5 X upper limit of normal (ULN)
  * Serum lipase >1.5 X ULN
  * Serum creatinine > 3.0 x ULN
* Subjects who have received an HIV prophylactic or corrective vaccination within 6 months prior to the first dose of study medication.
* Subjects who have received radiation therapy or cytotoxic chemotherapeutic agents and have not recovered from side effects prior to the first dose of study medication.
* Subjects with RT mutations Q151M or T69SS on Screening genotype.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with >= 1.0 log10 decrease in viral load from Baseline to Week 24 based on non-completer equals failure (NC=F) | Week 48 compared to baseline
Percent of subjects at 48 weeks with sustained suppression of viral load >= 1.0 log10 below baseline as determined by time-to-loss of virological response (TLOVR) | Week 48 compared to baseline

SECONDARY OUTCOMES:
Median change in viral load from Baseline to Week 24 and to Week 48 | Week 24 or Week 48 compared to baseline
Proportion of subjects in each treatment arm with viral load reduction greater than the over all study median viral load reduction | Week 24 and Week 48
Proportion of subjects with a viral load measurement <400 copies/mL at Week 24 and Week 48 | Week 24 and Week 48 compared to baseline
Proportion of subjects with a viral load measurement <50 copies/mL at Week 24 and Week 48 | Week 24 and Week 48 compared to Baseline
Median change in subset of T lymphocytes (CD4+) cell count from Baseline to Week 24 and Week 48 | Week 24 and Week 48 compared to baseline
Proportion of subjects with a 50% decrease and/or 100 cell/mm3 decrease in CD4+ cell count to Week 24 and to Week 48 | Week 24 and Week 48 compared to baseline
Proportion of subjects who "crossed-over" to receive treatment with the other blinded study medication | Week 16 and visits thereafter
Number of Centers for Disease Control (CDC) Class C adverse events and deaths by treatment arm | approximately every 2 to 4 weeks for laboratory testing

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Long Beach, California
  - Brandon, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Plantation, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - New York, New York
  - Portland, Oregon
  - Dallas, Texas
- San Juan, Puerto Rico